CLINICAL TRIAL: NCT07192692
Title: A Phase I Clinical Study to Evaluate the Effect of Food on the Pharmacokinetics of HSK47388 Tablets in Healthy Adult Subjects
Brief Title: Food Effect Study of HSK47388 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSK47388-104
Record Dates: First submitted 2025-08-28; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Pharmaceutical Preparations; Health Adult Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fast (Experimental): fast state
  Interventions: Dietary Supplement: fast
- low fat meal (Experimental): take HSK47388 with low fat meal
  Interventions: Dietary Supplement: low fat meal
- take meal after HSK47388 administration (Experimental): take meal after HSK47388 administration at specific time
  Interventions: Dietary Supplement: take meal after HSK47388 administration

INTERVENTIONS:
Dietary Supplement: fast — fast state
  Arms: fast
Dietary Supplement: low fat meal — take HSK47388 with low fat meal
  Arms: low fat meal
Dietary Supplement: take meal after HSK47388 administration — take meal after HSK47388 administration at specific time
  Arms: take meal after HSK47388 administration

SUMMARY:
This is a Phase 1, open-label, randomized, three-period crossover trial study to evaluate the effect of food and dosing and meal timing intervals on the pharmacokinetics (PK) of HSK46575 in healthy adult participants ,with an exploratory assessment of excretion pathways and excretion rates. Safety and tolerability will also be evaluated.

DETAILED DESCRIPTION:
The study consists of 3 treatment sequences in a 3-period, crossover design. Approximately 15 healthy adult participants will be randomized 1:1:1 to one of the following sequences:

Sequence A: Participants will receive HSK47388 orally in the fasted state (condition 1), administrate HSK47388 immediately after low-fat meal (condition 2), administrate HSK47388 in the fasted state, followed by a standard meal speicific minutes later（condition 3）.

Sequence B: Participants will receive administrate HSK47388 immediately after low-fat meal (condition 2), administrate HSK47388 in the fasted state, followed by a standard meal speicific minutes later（condition 3），HSK47388 orally in the fasted state (condition 1).

Sequence C: Participants will receive HSK47388 in the fasted state, followed by a standard meal speicific minutes later（condition 3),HSK47388 orally in the fasted state (condition 1), administrate HSK47388 immediately after low-fat meal (condition 2) .

All participants will remain under clinical observation for safety monitoring and pharmacokinetic sampling throughout each period. Blood, urine and fecal samples will be collected at defined intervals for the analysis of HSK47388 and its metabolites.

Each participant's total study duration will be approximately 37 days, including screening, treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
2. Adult males and females between ≥ 18 and ≤ 55 years (inclusive) at Screening.
3. Able and willing to attend the necessary visits to the study site

Exclusion Criteria:

1. Participants with any disease history that may affect the safety evaluation or in vivo process of IP as judged by the PI or delegate, including central nervous, cardiovascular, digestive, respiratory, urinary, blood, immune and endocrine diseases. Participants with childhood asthma (resolved) can be included at the discretion of the PI.
2. Underlying physical or psychological medical condition that, in the opinion of the PI or delegate, would make the participant unlikely to comply with the protocol or complete the study per protocol.
3. Participants who may not be able to complete the study for other reasons, cannot comply with the requirements of the study, or are unsuitable to participate in the study as judged by the PI or delegate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | 5 days after every period dose
  The incidence, severity, and relationship to IP of AEs. Change from Baseline in clinical laboratory parameters (ie, hematology, serum chemistry, coagulation, and urinalysis parameters), physical examination findings, vital signs

SECONDARY OUTCOMES:
pharmacokinetics of HSK47388 | time after 5 days in each period
  PK parameters: Cmax (Peak Plasma Concentration)
pharmacokinetics of HSK47388 | time after 5 days in each period
  PK parameters:Area under the plasma concentration versus time curve (AUC)
culmulative excretion rate | 5 days after dose in each period
  urine and feces culmulative excretion rate

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
for data confidence